CLINICAL TRIAL: NCT03417557
Title: Clinical Validation Study of Biofinity Multifocal Toric Contact Lenses
Brief Title: Clinical Validation Study of Comfilcon A Multifocal Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CV-18-10
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: This will be, prospective, single-masked, randomized, bilateral, cross-over, non-dispensing study comparing the test lens against the control lens.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Comfilcon A lens (test) (Experimental): Subjects are randomized to wear comfilcon A lens for up to 3 hours, either as first or second lens during this cross over study.
  Interventions: Device: Comfilcon A lens (test)
- Omafilcon B Lens (control) (Active Comparator): Subjects are randomized to wear omafilcon B lens for up to 3 hours, either as first or second lens during this cross over study.
  Interventions: Device: Omafilcon B lens (control)

INTERVENTIONS:
Device: Comfilcon A lens (test) — contact lens
  Other Names: Biofinity multifocal toric Lens (test)
  Arms: Comfilcon A lens (test)
Device: Omafilcon B lens (control) — contact lens
  Other Names: Proclear multifocal toric lens (control)
  Arms: Omafilcon B Lens (control)

SUMMARY:
This is a study to evaluate the clinical performance and subjective acceptance of an investigational contact lens (test), compared to a marketed lens (control) in an in-office setting.

DETAILED DESCRIPTION:
This is a study to evaluate the clinical performance (including visual acuity, subjective assessments of visual performance, comfort ratings, vision preference and lens fit) of a comfilcon A investigational contact lens (test) compared to a control contact lens, in a non-dispensing setting. The main study hypothesis is the test contact lens will not be clinically inferior to the control lens.

ELIGIBILITY:
Inclusion Criteria:

* Has had a self-reported oculo-visual examination in the last two years.
* Is between ages 40-75 years, inclusive and has full legal capacity to volunteer.
* Has read and understood the information consent letter. Is willing and able to follow instructions and maintain the appointment schedule.
* Is able to participate in Parts A and B related to this work.
* Has a contact lens spherical prescription between +10.00 to 10.00D (inclusive).
* Has an Add component to their spectacle refraction (between +0.75 and +2.50DS).
* Has astigmatism between of -0.75 and -5.75DC (based on the calculated ocular refraction) in each eye.
* Is correctable to a visual acuity of 20/40 or better (in each eye) with their habitual vision correction or 20/25 best-corrected.
* Currently wears soft contact lenses.
* Has clear corneas and no active ocular disease.
* Has not worn lenses for at least 12 hours before the examination.

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Optics Research Lab (CORL) Indiana University School of Optometry, Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three subjects did not meet the inclusion criteria. Seventeen (17) subjects completed all visits and were included in the analysis.
Groups:
- Comfilcon A Lens Then Omafilcon B Lens: Subjects are randomized to wear comfilcon A lens for up to 3 hours then omafilcon B lens for up to 3 hours during this cross over study.
  Comfilcon A lens (test): contact lens
- Omafilcon B Lens Then Comfilcon A: Subjects are randomized to wear omafilcon B lens for up to 3 hours then comfilcon A lens up to 3 hours during this cross over study.
  Omafilcon B lens (control): contact lens
Period: 1st Intervention (3 Hours)
Arm/Group | Comfilcon A Lens Then Omafilcon B Lens | Omafilcon B Lens Then Comfilcon A
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: 2nd Intervention (3 Hours)
Arm/Group | Comfilcon A Lens Then Omafilcon B Lens | Omafilcon B Lens Then Comfilcon A
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Comfilcon A Lens (Test) and Omafilcon B (Control): Subjects were randomized to wear the comfilcon A (test) or omafilcon B (control) lens for up to 3 hours, either as first or second lens during this cross over study.
Arm/Group | Comfilcon A Lens (Test) and Omafilcon B (Control)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual acuity is assessed for test and control lens on a logMAR chart
Time Frame: up to 3 hours
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Comfilcon A Lens (Test): Subjects are randomized to wear comfilcon A lens for up to 3 hours during this cross over study.
  Comfilcon A lens (test): contact lens
- Omafilcon B Lens (Control): Subjects are randomized to wear omafilcon B lens for up to 3 hours during this cross over study.
  Omafilcon B lens (control): contact lens
Arm/Group | Comfilcon A Lens (Test) | Omafilcon B Lens (Control)
Number analyzed (Participants) | 17 | 17
logMAR
  Distance: Binocular | -0.01 (0.09) | -0.03 (0.16)
  Distance: Monocular (dominate eye) | -0.05 (0.12) | 0.06 (0.21)
  Distant: Monocular (non-dominate eye) | 0.02 (0.13) | 0.13 (0.22)
  Near: Binocular | 0.05 (0.09) | 0.03 (0.07)
  Near: Monocular (dominate eye) | 0.14 (0.11) | 0.17 (0.13)
  Near: Monocular (non-dominate eye) | 0.10 (0.13) | 0.04 (0.18)

2. Secondary Outcome: Subjective Assessment of Visual Performance: Distance Day-time Navigation Tasks for Vision Quality and Clarity
Description: Subjective assessment of visual performance for distance day-time navigation tasks for vision/clarity was assessed for test and control lens at different testing distances. Scale 0-100, 0=poor, 100=excellent.
Time Frame: up to 3 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Lens (Test) | Omafilcon B Lens (Control)
Number analyzed (Participants) | 17 | 17
units on a scale | 91 (8) | 79 (24)

3. Secondary Outcome: Subjective Assessment of Visual Performance: Intermediate / Computer Task for Vision Quality and Clarity
Description: Subjective assessments of visual performance for intermediate / computer tasks for vision quality and clarity were assessed for test and control lens at different testing distances. Scale 0-100, 0=poor, 100=excellent.
Time Frame: up to 3 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Lens (Test) | Omafilcon B Lens (Control)
Number analyzed (Participants) | 17 | 17
units on a scale | 87 (12) | 82 (17)

4. Secondary Outcome: Subjective Assessment of Visual Performance: Near Vision for Vision Quality and Clarity
Description: Subjective assessments of visual performance for near vision was assessed for vision quality and clarity for test and control lens at different testing distances. Scale 0-100, 0=poor, 100=excellent.
Time Frame: up to 3 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Lens (Test) | Omafilcon B Lens (Control)
Number analyzed (Participants) | 17 | 17
units on a scale | 84 (17) | 79 (26)

ADVERSE EVENTS:
Time Frame: Up to 3 hours per intervention.
Arm/Group | Comfilcon A Lens (Test) | Omafilcon B Lens (Control)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT03417557/Prot_SAP_000.pdf